CLINICAL TRIAL: NCT05646420
Title: Deciphering the Role of Thyroid Hormones in Autosomal Dominant Polycystic Kidney Disease
Brief Title: Thyroid Hormones in ADPKD
Acronym: REORIENTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REORIENTED
Record Dates: First submitted 2022-12-05; First posted 2022-12-12 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Autosomal Dominant Polycystic Kidney
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADPKD patients (Experimental): The study will include 90 patients with diagnosis of ADPKD based on renal ultrasonography findings or genetic test.
  Specifically, five groups of patients will be identified according to KDIGO classification:
  * 18 subjects with normal or high renal function: eGFR ≥90 ml/min/1.73m2 - CKD G1 stage
  * 18 subjects with mildly decreased renal function: eGFR 89-60 ml/min/1.73m2 - CKD G2 stage
  * 18 subjects with mildly to moderately decreased renal function: eGFR 59 to 45 ml/min/1.73m2 - CKD G3a stage
  * 18 subjects with moderately to severely decreased renal function: eGFR 44 to 30 ml/min/1.73m2 - CKD G3b stage
  * 18 subjects with severely decreased renal function: eGFR 29 to 15 ml/min/1.73m2 - CKD G4 stage.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — A blood sample of 15 ml will be collected for each patient.

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is a monogenic, rare and life-threatening disease, characterized by the pathological formation of multiple fluid-filled cysts that arise from renal tubules and alter kidney architecture and function. In most patients, the progressive deterioration of renal function ultimately leads to end-stage kidney disease (ESKD) and the need for dialysis or kidney transplantation.

Save the conventional anti-hypertensive strategies, there are currently two disease-specific treatments for ADPKD (Tolvaptan and Octreotide-LAR). However, these drugs are only available to patients at high risk of progression to ESKD, while a remarkable number of ADPKD patients progress to ESKD despite the treatments.

Cyst formation in ADPKD is determined by mutations in two genes encoding two transmembrane proteins: polycystin1 and polycystin2. The pathogenesis of the disease involves a series of phenotypic alterations, including the de-differentiation of epithelial cells, uncontrolled proliferation and abnormal secretion of fluids in the cysts, metabolic remodeling, all phenomena that lead to the progressive loss of renal structure and function . Therefore, to try to investigate the mechanisms of the disease, the investigators should go in search of pleiotropic molecules capable of simultaneously modulating structure, function and metabolism.

Research done so far suggests that thyroid hormones (TH) may also act as pleiotropic modulators in the patho-biology of ADPKD. TH signals play a crucial role in the regulation of cell de-differentiation and cell cycle reactivation, as well as in the metabolism and evolution of cardiac and renal diseases. Interestingly, changes in TH levels have been detected in approximately 80% of patients with chronic renal failure (CKD), whereas patients with ADPKD show a higher incidence of clinical and subclinical hypothyroidism. Despite these evidences, the ability of TH to modulate anti-cystogenic and renoprotective processes in ADPKD has not yet been studied.

The objective of this study is to determine the levels of THs in the serum of ADPKD patients with normal renal function and mild, moderate or severe renal dysfunction, and to correlate them with renal functional parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥18 years old;
2. Diagnosis of ADPKD based on renal ultrasonography or genetic test;
3. Written informed consent

Exclusion Criteria:

1. Diagnosis of Hashimoto's disease, hyperthyroidism or pituitary disease or any other condition undergoing levothyroxine replacement
2. Patient with hypothyroidism treated with drug therapy
3. Active treatment with Tolvaptan and/or Octreotide-LAR;
4. Regular treatment with amiodarone, lithium, interferon or immunosuppressive drugs including steroids;
5. Active malignancy or acute or chronic inflammatory disease, HIV;
6. Dialysis or kidney transplantation;
7. Diabetes mellitus;
8. Hypocaloric diet or current dietary approaches to obtain weight loss.
9. Legal incapacity or any evidence that the patient will not be able to understand the study aims and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Serum levels of total and free triiodothyronine (T3). | Once during the study.
Serum levels of total and free L-thyroxine (T4). | Once during the study.
Serum levels of total and free thyroid stimulating hormone (TSH). | Once during the study.
Serum levels of total and free reverse T3 (rT3). | Once during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No